CLINICAL TRIAL: NCT02090114
Title: A Phase II Study to Determine Sequential Response to Bipolar Androgen Therapy (BAT) Followed by Enzalutamide or Abiraterone Post-BAT in Men With Prostate Cancer Progressing on Combined Androgen Ablative Therapies
Brief Title: RE-sensitizing With Supraphysiologic Testosterone to Overcome REsistance (The RESTORE Study)
Acronym: Restore
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1416; NA_00093344 (Other: JHM IRB); 1R01CA184012-01 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-18 (Estimated); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Bipolar Androgen Therapy; Testosterone; Enzalutamide; Abiraterone; Androgen Ablative Therapies
MeSH Terms: conditions — Prostatic Neoplasms | interventions — testosterone 17 beta-cypionate; testosterone enanthate; Abiraterone Acetate; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort A:Post-enzalutamide (Experimental): Men with castration-resistant prostate cancer who have progressed on enzalutamide will be enrolled to this cohort. These patients will then receive intramuscular injections with testosterone cypionate 400 mg every 28 days or testosterone enanthate 400 mg every 28 days. Upon progression on testosterone cypionate or enanthate, men will be retreated with enzalutamide 160 mg by mouth daily.
  Interventions: Drug: Testosterone cypionate; Drug: Testosterone Enanthate; Drug: Enzalutamide
- Cohort B: Post-abiraterone (Experimental): Men with castration-resistant prostate cancer who have progressed on abiraterone will be enrolled to this cohort. These patients will then receive intramuscular injections with testosterone cypionate 400 mg every 28 days or testosterone enanthate 400 mg every 28 days. Upon progression on testosterone cypionate or enanthate, men will be retreated with abiraterone 1000 mg by mouth daily.
  Interventions: Drug: Testosterone cypionate; Drug: Testosterone Enanthate; Drug: Abiraterone acetate
- Cohort C: Castration Only (Experimental): Men with metastatic prostate cancer who have only received first line hormone therapy with LHRH agonist alone or LHRH agonist plus an anti-androgen. Patients who have developed castrate resistance to first line therapy and have then received second line hormone therapy of any kind (including flutamide, bicalutamide, nilutamide, ketoconazole, abiraterone, enzalutamide, ARN-509 and investigational anti-androgens) are not eligible for enrollment in this cohort.
  Interventions: Drug: Testosterone cypionate; Drug: Testosterone Enanthate
- Cohort D: Mutation (Experimental): Men with metastatic prostate cancer who have castrate resistant prostate cancer with inactivating somatic or germline mutations in the genes TP53, RB1 or PTEN identified using clinical grade sequencing of tumor tissue performed by qualified laboratory. Patients must have mutations in ≥2 of these genes to be eligible. Eligible patients must have progressed on first line hormone therapy with LHRH agonist alone and must have received at least one but not more than two second generation androgen ablative therapy (i.e. Abiraterone, Enzalutamide or Apalutamide).
  Interventions: Drug: Testosterone cypionate; Drug: Testosterone Enanthate

INTERVENTIONS:
Drug: Testosterone cypionate — DEPO-Testosterone Injection, for intramuscular injection, contains testosterone cypionate which is the oil-soluble of the androgenic hormone testosterone. Testosterone cypionate is a white or creamy white crystalline powder, odorless or nearly so and stable in air. DEPO-Testosterone Injection is available in two strengths, 100 mg/mL and 200 mg/mL testosterone cypionate and will be administered at 400mg IM every 28 days.
  Other Names: DEPO-Testosterone Injection
Drug: Testosterone Enanthate — Testosterone Enanthate Injection, for intramuscular injection, contains testosterone enanthate which is the oil-soluble ester of the androgenic hormone testosterone. Enanthate Injection is available as a colorless to pale yellow solution. Each mL contains 200 mg testosterone enanthate in sesame oil with 5 mg chlorobutanol as a preservative. Will be administered at 400mg IM every 28 days.
  Other Names: Delatestryl
Drug: Abiraterone acetate — Abiraterone is an inhibitor of CYP17 (17α-hydroxylase/C17,20-lyase). Each ZYTIGA tablet contains 250 mg of abiraterone acetate.
  Other Names: Zytiga
  Arms: Cohort B: Post-abiraterone
Drug: Enzalutamide — XTANDI is provided as liquid-filled soft gelatin capsules for oral administration. Each capsule contains 40 mg of enzalutamide as a solution in caprylocaproyl polyoxylglycerides.
  Other Names: Xtandi
  Arms: Cohort A:Post-enzalutamide

SUMMARY:
Single-arm, single site, open label study of the effects of parenteral testosterone followed by enzalutamide, abiraterone or castration-only therapy in men with metastatic CRPC who previously progressed on one of these forms of therapy. The study will enroll four cohorts of patients: men with metastatic CRPC who have progressed on enzalutamide (Cohort A; n=30); men with metastatic CRPC who have progressed on abiraterone acetate (Cohort B; n=30); men with metastatic CRPC who have progressed on first line castration-only therapy (Cohort C; n=30); men with metastatic CRPC with inactivating somatic or germline mutations in ≥2 of the genes TP53, PTEN, or RB1 (Cohort D; n=20).

DETAILED DESCRIPTION:
The trial will enroll up to 110 patients, 30 for each Cohorts A-C and 20 for Cohort D. Eligible patients will continue on androgen ablative therapy with LHRH agonist (i.e. Zoladex, Trelstar, Eligard or Lupron) if not surgically castrated to suppress endogenous testosterone production. Patients will also receive intramuscular injection with either testosterone cypionate or testosterone enanthate at a dose of 400 mg every 28 days. This dosing scheme was designed to produce rapidly fluctuating serum testosterone levels from the supraphysiologic to the near-castrate range (i.e. Bipolar Androgen Therapy [BAT]). Assessments for response to testosterone will be made approximately every 3 months. Upon displaying evidence of progression, patients will then go on to receive either abiraterone (Cohort B) or enzalutamide (Cohort A), whichever agent they had previously progressed on prior to study enrollment. Patients in Cohort C will remain on LHRH agonist therapy and receive no additional androgen ablative hormonal therapy while those in the mutation-positive Cohort D will receive enzalutamide regardless of prior therapy.

ELIGIBILITY:
Inclusion Criteria:

* Performance status ≤2
* Age ≥18 years
* Histologically-confirmed adenocarcinoma of the prostate
* Progressing on continuous androgen ablative therapy (either surgical castration or LHRH agonist).
* Documented castrate level of serum testosterone (<50 ng/dl).
* For Cohorts A and B, patients must have progressed on prior treatment with enzalutamide or abiraterone acetate + prednisone (by PSA criteria or radiographically).
* For castration-only Cohort C, patients must have developed castrate resistant prostate cancer after progressing on first line hormone therapy with either surgical castration or LHRH agonist or LHRH agonist plus an anti-androgen.
* For Cohort D patients must have inactivating somatic or germline mutations in ≥2 of the genes TP53, PTEN, RB1
* Patients progressing on LHRH agonist plus an anti-androgen as first line therapy must be off anti-androgen for 4 weeks prior to first treatment with testosterone.
* Patients with rising PSA on two successive measurements at least two weeks apart.
* For Cohort A (enzalutamide) and Cohort B (abiraterone acetate):

  * Prior treatment with up to 2 additional second line hormone therapies, including ketoconazole is allowed.
  * Patients who have progressed on both enzalutamide and abiraterone acetate are eligible and post-BAT will be retreated with the last second line agent they had received (e.g. patient receiving abiraterone then enzalutamide would receive retreatment with enzalutamide post-BAT).
  * Patients must be withdrawn from enzalutamide or abiraterone acetate for ≥ 4 weeks and have documented PSA increase after the withdrawal period.
  * Patients receiving prednisone in conjunction with abiraterone acetate must be weaned off prednisone prior to starting BAT.
* For Cohort C (castration-only):

  * Patients must continue on castrating therapy throughout BAT treatment.
  * No prior second line hormone treatment with flutamide, bicalutamide, nilutamide, enzalutamide, abiraterone, ketoconazole, ARN-509 or other investigational androgen ablative therapies is permitted for Cohort C.
* For Cohort D (mutation cohort):

  * Patients must continue on castrating therapy throughout BAT treatment.
  * Treatment with first-generation hormonal therapy (i.e. flutamide, bicalutamide, nilutamide), is allowed
  * Patient must have received at least one and not more than two second generation hormone therapies (i.e. enzalutamide, abiraterone, apalutamide).
* For Cohorts A-D, prior docetaxel for hormone-sensitive prostate cancer is permitted if ≤ 6 doses were given in conjunction with first-line androgen deprivation therapy and >12 months since last dose of docetaxel
* For Cohort D, one line of prior chemotherapy with docetaxel or cabazitaxel for metastatic castrate resistant prostate cancer is allowed
* Acceptable liver function:

  * Bilirubin < 2.5 times institutional upper limit of normal (ULN)
  * AST (SGOT) and ALT (SGPT) < 2.5 times ULN
* Acceptable renal function:

  -- Serum creatinine < 2.5 times ULN, OR
* Acceptable hematologic status:

  * Absolute neutrophil count (ANC) ≥ 1500 cells/mm3 (1.5 ×109/L)
  * Platelet count ≥ 100,000 platelet/mm3 (100 ×109/L)
  * Hemoglobin ≥ 9 g/dL.
* At least 4 weeks since prior surgery with full recovery (no persistent toxicity ≥ Grade 1).
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Pain due to metastatic prostate cancer requiring opioid analgesics.
* >5 sites of visceral disease in lung or liver (nonspecific lung nodules ≤1 cm in diameter are permitted).
* Prior treatment with docetaxel or cabazitaxel for metastatic castration-resistant prostate cancer is prohibited.
* Prior treatment with one line of chemotherapy for metastatic castration-resistant prostate cancer is allowed for Cohort D
* Requires urinary catheterization for voiding due to obstruction secondary to prostatic enlargement thought to be due to prostate cancer or benign prostatic hyperplasia
* Evidence of disease in sites or extent that, in the opinion of the investigator, would put the patient at risk from therapy with testosterone (e.g. femoral metastases with concern over fracture risk, spinal metastases with concern over spinal cord compression, lymph node disease with concern for ureteral obstruction).
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study.
* Active uncontrolled infection, including known history of AIDS or hepatitis B or C.
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule.
* Prior history of a thromboembolic event within the last two years and not currently on systemic anticoagulation.
* Hematocrit >50%, untreated severe obstructive sleep apnea, uncontrolled or poorly controlled heart failure [per Endocrine Society Clinical Practice Guidelines (67)].

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-08-25 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Denmeade, MD, Principal Investigator — Johns Hopkins School of Medicine - Sidney Kimmel Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Markowski MC, Wang H, Sullivan R, Rifkind I, Sinibaldi V, Schweizer MT, Teply BA, Ngomba N, Fu W, Carducci MA, Paller CJ, Marshall CH, Eisenberger MA, Luo J, Antonarakis ES, Denmeade SR. A Multicohort Open-label Phase II Trial of Bipolar Androgen Therapy in Men with Metastatic Castration-resistant Prostate Cancer (RESTORE): A Comparison of Post-abiraterone Versus Post-enzalutamide Cohorts. Eur Urol. 2021 May;79(5):692-699. doi: 10.1016/j.eururo.2020.06.042. Epub 2020 Jul 2. PMID 32624280
- [Result] Sena LA, Wang H, Lim ScM SJ, Rifkind I, Ngomba N, Isaacs JT, Luo J, Pratz C, Sinibaldi V, Carducci MA, Paller CJ, Eisenberger MA, Markowski MC, Antonarakis ES, Denmeade SR. Bipolar androgen therapy sensitizes castration-resistant prostate cancer to subsequent androgen receptor ablative therapy. Eur J Cancer. 2021 Feb;144:302-309. doi: 10.1016/j.ejca.2020.11.043. Epub 2020 Dec 29. PMID 33383350
- [Result] Teply BA, Wang H, Luber B, Sullivan R, Rifkind I, Bruns A, Spitz A, DeCarli M, Sinibaldi V, Pratz CF, Lu C, Silberstein JL, Luo J, Schweizer MT, Drake CG, Carducci MA, Paller CJ, Antonarakis ES, Eisenberger MA, Denmeade SR. Bipolar androgen therapy in men with metastatic castration-resistant prostate cancer after progression on enzalutamide: an open-label, phase 2, multicohort study. Lancet Oncol. 2018 Jan;19(1):76-86. doi: 10.1016/S1470-2045(17)30906-3. Epub 2017 Dec 14. PMID 29248236

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 patients failed screen.
Period: Overall Study
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Started | 30 | 29 | 29 | 8
Completed | 0 | 0 | 0 | 0
Not Completed | 30 | 29 | 29 | 8
Not completed — Withdrawal by Subject | 3 | 6 | 2 | 1
Not completed — Physician Decision | 5 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 2 | 2 | 0
Not completed — Progressive Disease | 20 | 21 | 23 | 6
Not completed — Death | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation | Total
Number analyzed (Participants) | 30 | 29 | 29 | 8 | 96
Age, Continuous [Median (Full Range); unit: Years] | 74 [50 to 89] | 71 [49 to 85] | 69 [41 to 84] | 73 [56 to 89] | 72 [41 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 30 | 29 | 29 | 8 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 26 | 24 | 7 | 81
  Unknown or Not Reported | 6 | 3 | 4 | 0 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27 | 26 | 23 | 7 | 83
  Non-white | 3 | 3 | 6 | 1 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 29 | 29 | 8 | 96

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response to Bipolar Androgen Therapy (BAT)
Description: Number of participants with ≥50% PSA reduction from pre-BAT baseline level
Time Frame: up to 18 months
Population: Only 7/8 patients were evaluable from Cohort D.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 30 | 29 | 29 | 7
Participants | 9 | 5 | 4 | 2

2. Primary Outcome: PSA Response to Enzalutamide or Abiraterone Acetate Post Bipolar Androgen Therapy
Description: Number of participants with ≥50% PSA reduction after enzalutamide or abiraterone acetate post-BAT from baseline
Time Frame: up to 24 months
Population: This outcome measure only applies to cohort A,B, and D. Only 22/30 (Cohort A), 19/29 (Cohort B) and 7/8 (Cohort D) patients had evaluable data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 22 | 19 | 0 | 7
Participants | 15 | 3 |  | 2

3. Secondary Outcome: PSA Progression on Enzalutamide or Abiraterone Acetate or Castrate Levels Post-BAT
Description: Time to PSA progression on enzalutamide or abiraterone acetate or return to castrate levels of testosterone post-BAT, defined as the time from the date of re-initiation of enzalutamide or abiraterone acetate or castration-only therapy to the date of the PSA measurement when it shows an increase by ≥25% above the nadir value that occurred following re-initiation of enzalutamide or abiraterone acetate or castration-only therapy and confirmed by a repeat PSA 4 weeks later (PCWG2).
Time Frame: up to 18 months
Population: Only 21/30 participants were evaluable from Cohort A. Only 19/29 participants were evaluable from Cohort B.This outcome measure does not apply to Cohort D.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 21 | 19 | 29 | 0
months | 5.5 [4.6 to NA] — insufficient number of participants with events | 3.7 [1.5 to 5] | NA [NA to NA] — insufficient number of participants with events |

4. Secondary Outcome: PSA Progression on BAT (Bipolar Androgen Therapy )
Description: Time to PSA progression on BAT. Time to PSA progression on BAT is defined as the time from the date of initial dose of Testosterone to the date of the PSA measurement when it shows an ≥25% increase above the nadir value and confirmed by a repeat PSA 4 weeks later (PCWG2 criteria) during the treatment with BAT.
Time Frame: up to 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 30 | 29 | 29 | 7
months | 3.3 [2.7 to 5.5] | 3.2 [2.5 to 6] | 0.93 [0.93 to 5.58] | 3 [2.8 to NA] — insufficient number of participants with events

5. Secondary Outcome: Disease Response as Defined by RECIST 1.1 (Soft Tissue Lesions) and PCWG2 Criteria (Bone Lesions)
Description: Number of participants with complete or partial response post-BAT as defined by RECIST 1.1 (for soft tissue lesions) and PCWG2 criteria (for bone disease), or return to castration-only post-BAT.
Time Frame: up to 18 months
Population: 12/30 participants from Cohort A, 7/29 participants from Cohort B, 13/20 from Cohort C, and 7/8 participants from Cohort D were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 12 | 7 | 13 | 7
Participants | 6 | 2 | 4 | 0

6. Secondary Outcome: Initiation of Docetaxel Chemotherapy
Description: Time to initiation of docetaxel chemotherapy
Time Frame: up to 18 months
Population: Data was not collected to assess this outcome measure.
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Quality of Life (QoL) as Assessed by FACIT-F Score
Description: Functional Assessment of Chronic Illness Therapy, Fatigue Subscale (FACIT-F) assesses Fatigue with a total score range of 0-52, with a higher score reflecting better QoL.
Time Frame: up to 18 months
Population: 25/30 participants in Cohort A, 22/29 participants in Cohort B, 28/29 participants in Cohort C were evaluable for this outcome measure. Data was not collected from participants for Cohort D.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 25 | 29 | 29 | 0
score on a scale
  Baseline: number analyzed (Participants) | 25 | 22 | 28 | 0
  Baseline | 13.28 (6.73) | 16.86 (7.62) | 13 (5.57) |
  Cycle 1 Day 85 | 10.64 (5.51) | 13.85 (7.42) | 11.55 (3.39) |

8. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Adverse Events
Description: Number of participants who experience adverse events, as defined by NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: 18 months
Population: In cohort D, data was only collected from 7/8 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 30 | 29 | 29 | 7
Participants | 30 | 29 | 29 | 7

9. Secondary Outcome: Quality of Life (QoL) as Assessed by RANDSF-36
Description: RAND 36-Item Short Form (RANDSF-36) assesses physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, general health perceptions, and perceived change in health with a total score range of 0-100. The total score from all of the questions answered is divided by the total number of the questions answered yielding a global score from 0-100, with a higher score reflecting a better QoL.
Time Frame: up to 18 months
Population: 25/30 participants in Cohort A, 19/29 participants in Cohort B, 25/29 participants in Cohort C were evaluable for this outcome measure. Data was not collected from participants in Cohort D.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 30 | 29 | 29 | 0
score on a scale
  Baseline: number analyzed (Participants) | 25 | 19 | 25 | 0
  Baseline | 72.23 (18.89) | 64.36 (18.70) | 69.72 (17.72) |
  Cycle 1 Day 85 | 71.76 (19.20) | 73.97 (19.96) | 73.40 (17.98) |

10. Secondary Outcome: Quality of Life (QoL) as Assessed by BPI
Description: Brief Pain Inventory (BPI) assesses the severity of pain and its impact on functioning with scales ranging from 0-10, with a higher score indicating a higher level of pain.
Time Frame: up to 18 months
Population: Data was not collected for this outcome measure.
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Quality of Life (QoL) as Assessed by IIEF
Description: International Index of Erectile Function (IIEF-5) is a diagnostic tool for erectile dysfunction, with a total score range of 5-25, with the lowest score indicating a higher degree of dysfunction.
Time Frame: up to 18 months
Population: 20/30 participants in Cohort A, 21/29 participants in Cohort B, 25/29 participants in Cohort C were evaluable for this outcome measure. Data was not collected from participants in Cohort D.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 30 | 29 | 29 | 0
score on a scale
  Baseline | 8 (3.57) | 7.33 (3.89) | 12.56 (12.86) |
  BAT C1D85 | 24.13 (21.63) | 24.94 (19.71) | 22.44 (15.53) |

12. Secondary Outcome: Quality of Life (QoL) as Assessed by PANAS
Description: Positive and Negative Affect Schedule (PANAS) is a self-report measure that is made up of two mood scales, one measuring positive affect and the other measuring negative affect, with a total score range from 10-50 with a higher score on the positive scale indicating greater levels of positive affect and a lower score on the negative scale indicating less of a negative affect.
Time Frame: up to 18 months
Population: 20/30 participants in Cohort A, 18/29 participants in Cohort B, 25/29 participants in Cohort C were evaluable for this outcome measure. Data was not collected for Cohort D.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
Number analyzed (Participants) | 30 | 29 | 29 | 0
score on a scale
  Baseline: number analyzed (Participants) | 20 | 18 | 25 | 0
  Baseline | 46.15 (10.55) | 48 (11.47) | 41.24 (14.35) |
  BAT C1D85 | 45.1 (9.09) | 45.22 (12.94) | 44.48 (11.06) |

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Cohort A:Post-enzalutamide | Cohort B: Post-abiraterone | Cohort C: Castration Only | Cohort D: Mutation
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/29 | 1/29 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/30 | 4/29 | 5/29 | 1/8
Other Adverse Events (participants affected / at risk) | 30/30 | 29/29 | 29/29 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A:Post-enzalutamide (N=30) | Cohort B: Post-abiraterone (N=29) | Cohort C: Castration Only (N=29) | Cohort D: Mutation (N=8)
Urine Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis, elevated lipase, amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurological Symptoms (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A:Post-enzalutamide (N=30) | Cohort B: Post-abiraterone (N=29) | Cohort C: Castration Only (N=29) | Cohort D: Mutation (N=8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (39) | 8 (23) | 11 (22) | 4 (7)
Increased Hemoglobin (Blood and lymphatic system disorders) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 7 (24) | 4 (8) | 6 (6) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (16) | 7 (10) | 0 (0) | 2 (2)
Breast Tenderness (Reproductive system and breast disorders) | 5 (5) | 5 (6) | 6 (6) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (2) | 0 (0) | 0 (0)
fatigue (General disorders) | 17 (23) | 5 (5) | 5 (5) | 0 (0)
nausea (Gastrointestinal disorders) | 7 (9) | 4 (4) | 1 (1) | 1 (1)
gynecomastia (Reproductive system and breast disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
hot flashes (Vascular disorders) | 5 (6) | 4 (4) | 2 (4) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
edema (General disorders) | 4 (5) | 8 (12) | 7 (8) | 1 (3)
fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
sinusitis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
gallstone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 3 (3) | 5 (7) | 1 (1) | 1 (1)
headache (Nervous system disorders) | 3 (3) | 5 (5) | 1 (1) | 0 (0)
elevated ALK Phos (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
pain at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 2 | 1 (1) | 0 (0)
urine obstruction (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
increased hair growth (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
polycythemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
fever (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
constipation (Gastrointestinal disorders) | 3 (3) | 3 (4) | 1 (1) | 1 (2)
bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
weight loss (Investigations) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (6) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
chest pain (General disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Taster change (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine Increased (Investigations) | 3 (4) | 1 (1) | 1 (2) | 1 (1)
cold symptoms (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
High cholesterol (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Elevated potassium (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated hematocrit (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated Glucose (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated liver enzymes (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated AST (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated troponin (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
eye discorder (Eye disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT02090114/Prot_SAP_000.pdf